CLINICAL TRIAL: NCT00869505
Title: A Chart Review of Memantine Use in the Treatment of Obsessive-Compulsive Disorder at the OCD Institute
Brief Title: Study of Memantine Augmentation in Severe Obsessive-Compulsive Disorder
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: OCD Institute (Unknown); Mclean Hospital (Other)
Responsible Party: S. Evelyn Stewart, M.D., Director of Research, OCD Institute, Harvard Medical School, Massachusetts General Hospital, McLean Hospital
Other Study IDs: 2008-P-000461
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2009-03-26 (Estimated); Status verified 2009-03

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: To evaluate the effectiveness of memantine as an augmenting agent for standard intensive residential treatment of severe obsessive-compulsive disorder (OCD)
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case Group: Intensive Residential Treatment with memantine augmentation
- Control Group: Intensive Residential Treatment without memantine augmentation

SUMMARY:
Memantine is a glutamate receptor antagonist that has been reported to reduce Obsessive-Compulsive Disorder (OCD) symptoms in case studies of treatment-resistant individuals. The investigators hypothesized that memantine is an effective augmenting agent to standard intensive residential treatment of severe OCD. An intent-to-treat, single-blinded, naturalistic case-control design is employed. The sample includes subjects receiving standard treatment at the McLean/ MGH Intensive Residential Treatment (IRT) program, half of whom also receive memantine augmentation. Admission, monthly and discharge measures of OCD, depression and psychosocial functioning are collected by raters blinded to augmentation status. Matched controls are selected based upon gender, initial OCD severity, psychosocial functioning, and timing of admission. Descriptive and comparative analyses are conducted via SPSS, statistical significance is defined at p<0.05, clinically significant response is defined by a 25% reduction, and 'marked response' is defined by a 50% improvement in Yale-Brown Obsessive Compulsive severity (Y-BOCS) scores, using a last-observation-carried-forward approach. The Clinical Global Improvement (CGI) scale captures global clinical change.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients of IRT at the OCD Institute who agreed to augmentation with memantine.
* Consecutive patients of IRT at the OCD Institute who were not offered augmentation with memantine and who were matched according to OCD severity, gender, and psychosocial functioning.

Exclusion Criteria:

* Subjects offered memantine augmentation who did not provide voluntary consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprised 44 subjects who received standard treatment at the MGH/ McLean Hospital OCD Institute Intensive Residential Treatment (IRT) program, admitted between May 1999 and December 2007.
Sampling Method: Non-Probability Sample
Dates: Start 2008-03

CONTACTS AND LOCATIONS:
Overall Officials: S. Evelyn Stewart, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- OCD Institute, McLean Hospital, Belmont, Massachusetts, United States